CLINICAL TRIAL: NCT03847285
Title: Immune Function as Predictor of Infectious Complications and Clinical Outcome in Patients Undergoing Solid Organ Transplantation: A Prospective Non-interventional Observational Trial
Brief Title: Immune Function as Predictor of Infectious Complications and Clinical Outcome in Patients Undergoing Solid Organ Transplantation
Acronym: Immune-Mo
Status: Active, not recruiting | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Susanne Dam Nielsen, MD, DMSc, Principal investigator, clinical professor, Rigshospitalet, Denmark
Other Study IDs: sponsor - rigshospitalet
Record Dates: First submitted 2019-02-06; First posted 2019-02-20 (Actual); Last update posted 2024-04-10 (Actual); Status verified 2024-04

CONDITIONS: Transplant
Keywords: Transplant; Infection; rejection; immunology
MeSH Terms: conditions — Infections; Rejection, Psychology

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — whole blood and plasma
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: solid organ transplantation — solid organ transplantation: kidney, heart, pancreas, lung and liver transplantation

SUMMARY:
At Rigshospitalet, Denmark, we will examine the immune function of solid organ transplant recipients before and at several timepoints after transplantation as well as the clinical outcome, especially the risk of infections complications and graft rejections.

The immune function will be assessed with a complete immunological profiling consisting of immune phenotype (flow cytometry), immune function (TruCulture®) and circulating biomarkers.

The study aims to generate prediction models of patients at excess risk of poor clinical outcome, with the ultimate intent to propose personalized immunosuppressive regimes to be tested in future randomized clinical trials.

DETAILED DESCRIPTION:
Background: Solid organ transplantation (SOT) is an increasingly used life-saving treatment for end-stage organ failure. Organ rejection and infections are the main complication to SOT and the balance of immunosuppression is of major importance to prevent these complications. However, to date the only mode to monitor treatment is by assessing drug concentrations, which has low correlation with the clinical outcome and does not represent the net state of immunosuppression.

Methods: Prospectively the investigators plan to enroll 600 adult patients on the waiting list for SOT or with a planned transplantation at Rigshospitalet, Denmark. Prior to transplantation and on different time points up to two years post-transplantation we will perform a complete immunological profile. This profile will consist of classical descriptive immune phenotyping (flowcytometry), circulating biomarkers and the functional assay TruCulture®. In TruCulture® whole blood is stimulated with stimulants imitating bacterial, viral and fungal infections, where after a panel of selected cytokines is quantified.

Clinical data from electronic health records will be obtained retrospectively from the PERSIMUNE data repository. These data are generated as part of routine care and include vital signs, biochemistry-, microbiological-, pathological-results as well as data about medication, demographics, diagnoses, hospital contacts, surgical procedures and mortality.

Discussion: This will be the first large scale study to determine several aspects of immune function and perform a complete immunological profiling in SOT recipients. It is expected that this new knowledge will provide information to generate prediction models identifying patients at increased risk of infection and/or rejection. If the study is successful, the investigators will subsequently use the generated prediction models to propose personalized immunosuppressive regimens to be tested in future randomized controlled trials.

ELIGIBILITY:
Inclusion Criteria:

* To be eligible for the study the participant must be a minimum of 18 years of age, participate in the PERSIMUNE biobank, have a planned kidney, heart, lung, liver or pancreas transplant or be on the waiting list for a heart, lung, liver or pancreas transplant and be able to sufficiently understand oral and written study information in Danish or English to provide an informed consent. Study participation is strictly voluntary

Exclusion Criteria:

* not meeting inclusion criteria

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Participants must have a planned kidney, heart, lung, liver or pancreas transplant or be on the waiting list for a heart, lung, liver or pancreas-transplantation at Rigshospitalet, Denmark
Sampling Method: Non-Probability Sample
Enrollment: 188 (Actual)
Dates: Start 2018-04-01 (Actual); Primary Completion 2022-01-31 (Actual); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Infection | one year
  Infections (viral, bacterial or fungal) within 1 year after the transplantation
graft rejection | one year
  Graft rejection within 1 year after the transplantation. Rejections will be defined by pathologist and clinician.

SECONDARY OUTCOMES:
combined endpoints at 28 days post transplantation | 28 days
  Combined endpoint of infections (viral, bacterial or fungal) or graft rejection within 28 days
combined endpoints at 90 days post transplantation | 90 days
  Combined endpoint of infections (viral, bacterial or fungal) or graft rejection within 90 days
combined endpoints at 2 years post transplantation | 2 years
  Combined endpoint of infections (viral, bacterial or fungal) or graft rejection within 2 years
combined endpoints at 5 years post transplantation | 5 years
  Combined endpoint of infections (viral, bacterial or fungal) or graft rejection within 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Susanne Dam Nielsen, DMSc, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Drabe CH, Sorensen SS, Rasmussen A, Perch M, Gustafsson F, Rezahosseini O, Lundgren JD, Ostrowski SR, Nielsen SD. Immune function as predictor of infectious complications and clinical outcome in patients undergoing solid organ transplantation (the ImmuneMo:SOT study): a prospective non-interventional observational trial. BMC Infect Dis. 2019 Jul 3;19(1):573. doi: 10.1186/s12879-019-4207-9. PMID 31269923